CLINICAL TRIAL: NCT00708851
Title: A Clinical Evaluation of Safety & Efficacy of Adding an At-home Topical LCD Solution Regimen to Standard Narrowband UVB Phototherapy Administered 3 Times Weekly to Adults With Generalized Plaque Psoriasis.
Brief Title: NB-UVB Phototherapy With and Without Topical LCD Treatment: a Bilateral Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoStrata Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 07-LCDUVB
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB-UVB Light Device (311-315 nm) (Active Comparator): the subject will receive full body NB-UVB light therapy
  Interventions: Device: NB-UVB Light Device (311-315 nm)
- LCD Solution with NB-UVB Phototherapy (Experimental): on half of the body will receive LCD while the full body receives NB-UVB therapy
  Interventions: Other: LCD Solution with NB-UVB Phototherapy; Device: NB-UVB Light Device (311-315 nm)

INTERVENTIONS:
Other: LCD Solution with NB-UVB Phototherapy — LCD Solution: 2 applications / day
  NB-UVB Phototherapy: 3 light sessions / week
  Other Names: LCD
  Arms: LCD Solution with NB-UVB Phototherapy
Device: NB-UVB Light Device (311-315 nm) — NB-UVB Phototherapy: 3 light exposures / week
  Other Names: Ultralite Model # V4848NB

SUMMARY:
The purpose of this study is to determine if combining a daily at-home regimen using an LCD Solution with a 3 times weekly outpatient narrowband UVB phototherapy regimen could be a safe, effective, rapid, and, convenient treatment for plaque psoriasis.

DETAILED DESCRIPTION:
Use of coal tar with narrowband (NB) ultraviolet B (UVB) light (the Goeckermen regimen) is an effective treatment for plaque psoriasis that has become impractical in outpatient care mainly due to the inconvenience and aesthetic concerns of coal tar. This study aims to evaluate the safety, efficacy, and convenience of adding a novel liquor carbonis distillate (LCD) (coal tar) solution to standard NB_UVB phototherapy in adults with chronic plaque psoriasis. Patients will apply LCD solution to half the body, twice daily at home and receive outpatient full-body NB-UVB light therapy 3 times a week for up to 12 weeks. A blinded investigator will grade psoriasis severity of body halves and bilateral target lesions and monitor adverse reactions. Patients will rate their psoriasis symptoms and LCD solution aesthetics. Incorporating an at-home regimen with a novel LCD solution into outpatient NB-UVB light therapy is safe, convenient, and effective and can improve psoriasis more quickly than NB-UVB light therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* able and willing to provide written informed consent
* symmetrical plaque psoriasis
* able and willing to attend phototherapy sessions and apply LCD at home
* negative pregnancy test for women of child-bearing potential

Exclusion Criteria:

* current or recent other treatments for psoriasis
* hypersensitivity to LCD or UVB light
* current or previous skin cancer
* pregnant or nursing mother
* participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Bagel, MD, Principal Investigator — Windsor Dermatology, East Windsor, NJ 08520
Locations (1):
- Windsor Dermatology, East Windsor, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NB-UVB and NB-UVB+LCD: NB-UVB Alone: NB-UVB Light Device (311-315 nm) NB-UVB Phototherapy: 3 light exposures / week
  NB-UVB+LCD: 2 applications of LCD/day + NB-UVB Light Device (311-315 nm): NB-UVB Phototherapy 3 light exposures / week
Period: Overall Study
Arm/Group | NB-UVB and NB-UVB+LCD
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 12 participants with bilateral, symmetrical plaque psorasis
Groups:
- NB-UVB Alone: One leg receives NB-UVB Alone: NB-UVB Light Device (311-315 nm): NB-UVB Phototherapy: 3 light exposures / week
  Opposite leg receives: LCD therapy 2 applications/day and NB-UVB Light Device (311-315 nm) NB-UVB Phototherapy 3 light exposures / week
Arm/Group | NB-UVB Alone
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 44.41 [25 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Bilateral Static Physician's Global Assessment (sPGA) Scores, and Erythema, Scaling, and Induration (ESI) Scores of Bilateral Target Lesion Scores Across Visits for Each Condition and Between Conditions.
Description: Twelve (12) participants were followed over a 12-week treatment period. Treatment was administered bilaterally as they applied LCD solution to one half of their body while receiving full-body NB-UVB light therapy. The difference in their sPGA, and ESI scores of bilateral target lesions were measured across all visits. PGA scores are calculated using a 6-point scale from 0 (clear) to 5 (very severe). Erythema, induration and scaling scores use a 5-point scale from 0 (none) to 4 (very severe).
Time Frame: 12 weeks of treatment
Population: Data were analyzed using an intent-to-treat (ITT) population. All enrolled patients were included in the analysis. Missing scores we filled in by last observation carried forward method. All statistical tests were two-sided and used a level of significance of alpha = 0.05.
Measure: Mean (Full Range); unit: percent improvement from baseline
Groups:
- NB-UVB Alone: NB-UVB Alone
  NB-UVB Light Device (311-315 nm): NB-UVB Phototherapy: 3 light exposures / week
- LCD+NB-UVB: LCD+NB-UVB
  LCD Solution with NB-UVB Phototherapy: LCD Solution: 2 applications / day
  NB-UVB Phototherapy: 3 light sessions / week
Arm/Group | NB-UVB Alone | LCD+NB-UVB
Number analyzed (Participants) | 12 | 12
percent improvement from baseline
  Percent Change in PGA score from Baseline | 77.8 [0 to 100] | 85.4 [1 to 100]
  Mean Percent Change in Erythema | 88.5 [0 to 100] | 88.9 [0 to 100]
  Mean Percent Change in Induration | 84.2 [0 to 100] | 85.7 [0 to 100]
  Mean Percent Decrease in Desquamation | 65.2 [0 to 100] | 82.6 [0 to 100]

2. Secondary Outcome: The Difference in Number and Severity of Treatment-related Adverse Reactions Between Conditions.
Description: Number of subjects who experienced and adverse reaction due to UVB + LCD, versus number of subjects who experienced an adverse reaction due to UVB therapy alone.
Time Frame: 12 weeks of treatment
Population: Data were analyzed using an intent-to-treat (ITT) population. All enrolled patients were included in the analysis. Missing scores were filled in by last observation carried forward method. All statistical tests were two-sided and used a level of significance of alpha = 0.05.
Measure: Number; unit: participants
Arm/Group | NB-UVB Alone | LCD+NB-UVB
Number analyzed (Participants) | 12 | 12
participants | 3 | 3

ADVERSE EVENTS:
Time Frame: Adverse events for this study were monitored and documented throughout the entire 12 week study.
Description: Adverse events were reported directly by the subject to the principal investigator, who then informed the responsible party: NeoStrata Co., Inc.
Arm/Group | NB-UVB Alone | LCD+NB-UVB
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NB-UVB Alone (N=12) | LCD+NB-UVB (N=12)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — adverse reaction consisted of one report of mild post-NB-UVB erythema, which appeared uniformly on both sides of the body, regardless of treatment condition.
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Treatment-related adverse reactions consisted of two reports of moderate post-UVB erythema which appeared uniformly on both sides of the body.

LIMITATIONS AND CAVEATS:
This is a bilateral pilot study including 12 subjects. Subjects will apply the liquor carbonis distillate (LCD) solution to one half of their body, while receiving narrow-band ultraviolet B (NB-UVB) light therapy across their whole body.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No